CLINICAL TRIAL: NCT02522520
Title: Pedometer Intervention, Health Counseling, Symptom Management for Sedentary Colorectal Cancer Patients During Adjuvant Chemotherapy.Two-armed Randomized Phase II Trial
Brief Title: Pedometer Intervention and Health Effects for Sedentary Colorectal Cancer Patients During Adjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Novo Nordisk A/S (Industry); Danish Cancer Society (Other); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Christina Andersen, RN, MPH, Ph.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CIRE-15
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
Keywords: Undergoing chemotherapy; Exercise intervention; Health counselling; Symptom management
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcome (VO2 peak) Physiological tests assessors blinded
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pedometer intervention (Active Comparator): Individual progressive pedometer intervention of low to moderate intensity.
  Furthermore, the patients receive individual health counseling and symptom management counseling to support behavioral change towards increased physical activity.
  Interventions: Behavioral: Pedometer intervention; Device: Omron Walking Style pro. 20
- Pedometer + hospital based intervention (Active Comparator): Individual progressive pedometer intervention and 5 sessions supervised interval walking + followed by supervised hospital-based intervention of moderate to high-intensity
  Furthermore, the patients receive individual health counseling and symptom management counseling to support behavioral change towards increased physical activity.
  Interventions: Behavioral: Pedometer + hospital based intervention; Device: Omron Walking Style pro. 20

INTERVENTIONS:
Behavioral: Pedometer intervention — 12 weeks physical activity intervention (supervised/non-supervised)
  Arms: Pedometer intervention
Behavioral: Pedometer + hospital based intervention — 12 weeks physical activity intervention (supervised/non-supervised)
  Arms: Pedometer + hospital based intervention
Device: Omron Walking Style pro. 20
  Other Names: Pedometer

SUMMARY:
Colorectal cancer is one of the most common cancers in Denmark, annually 4,200 men and women are diagnosed and approx. 2000 patients die of their colorectal cancer. As with other cancers, the risk of colorectal cancer increases with age, and the median age at diagnosis is 71 years. Improved treatment has increased the number of survivors with an expected 5-year survival rate of 50-60%. Characteristic of this group of patients is that at the time of diagnosis they often live with comorbidities and have limited leisure time physical activity.

There is evidence that rehabilitation in the form of physical exercise for cancer patients after their initial treatment has a positive effect on a number of physical and psychological parameter such as health-related quality of life, physical capacity and physical function, fatigue, anxiety and depression. However, the most frequently studied diagnosis group is women with breast cancer. Until now only few studies have evaluated the effects of physical activity among colorectal cancer patients receiving chemotherapy

The purpose of this study is: to examine the effect of two different training initiatives - 12 weeks progressive, high-intensity training versus low intensity exercise intervention - on physical, emotional and social habitus, in sedentary patients with colorectal cancer during adjuvant chemotherapy.

The hypothesis of the study are: 1. That both interventions will show a positive association between increased physical capacity (measured by aerobic capacity VO2-peak / peak oxygen uptake) and improved physical function, reduced fatigue and anxiety in the included sedentary colorectal cancer patients undergoing adjuvant chemotherapy.

Participants: Patients undergoing adjuvant chemotherapy for colorectal cancer who have self-reported physical activity level below the national recommended levels (less than 150 min/week of moderate leisure time physical activity, and exercises at least 20 minutes of strenuous physical activity twice a week).

Benefits and risks of participating: Possible benefits of the interventions: to reduce treatment related symptoms and side-effects, increase vitality and well-being and promote lifestyle changes among sedentary colorectal cancer patients receiving adjuvant chemotherapy. At participation in the interventions minor sports injuries may occur.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal cancer in adjuvant chemotherapy
* Age 18+ years
* WHO performance status of 0 or 1
* Undergone surgery at least 6 weeks ago
* Do not meet criteria for recommended physical activity level of 150 min / week of moderate leisure time physical activity, and exercises at least 20 minutes of strenuous physical activity twice a week.

Exclusion Criteria:

* Myocardial infarction within the past six months
* Symptomatic heart failure
* Known angina pectoris
* Contraindication for moderate to strenuous physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2020-06 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen uptake - ( VO2 peak) | 12 weeks
  Assessed with objective physiological test

SECONDARY OUTCOMES:
Health related Quality of Life | From baseline to 39 weeks
  Assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, specifically for colon cancer patients
Symptoms and side-effects | From baseline to 39 weeks
  Assessed by MD Andersen symptom questionnaire and The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, chemotherapy-induced peripheral neuropathy
Anxiety and Depression | From baseline to 39 weeks
  Assessed by The Hospital Anxiety and Depression Scale
Lifestyle factors | From baseline to 39 weeks
  Assessed by smoking cessation, alcohol, diet
Physical activity level | From baseline to 39 weeks
  Assessed by the International Physical Activity Questionnaire
Dual Energy X-ray Absorptiometry scan | From baseline to 39 weeks
  Assessed by dual energy x-ray absorptiometry.
Blood cholesterols | From baseline to 39 weeks
  Assessed by blood samples
Blood pressure / pulse | From 6 to 12 weeks
  Assessed by Heart Rate Monitor during the hospital-based intervention
Pedometer Step Count | From baseline to 12 weeks
  Assessed by Omron Walking Style pro. 20 with electronic data transmission

CONTACTS AND LOCATIONS:
Overall Officials: Lis Adamsen, Professor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Presently no plan to make IPD available to other researchers